CLINICAL TRIAL: NCT05394584
Title: The Implementation of Cognitive Stimulation Therapy Hong Kong Version (CST-HK) for Promoting Cognitive Functioning and Psychosocial Well-being of People With Dementia
Brief Title: CST-HK for Cognition and Well-being in People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Young Women's Christian Association (Other); Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA1802054
Record Dates: First submitted 2022-05-17; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Dementia of Alzheimer Type
Keywords: Cognitive Stimulation Therapy; Cognitive Functioning; Psychological Wellbeing

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized wait-list control study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CST group (Experimental): A total of 64 people with mild-to-moderate cognitive impairment will receive group cognitive stimulation therapy (CST), which consists of 14 sessions of mentally stimulating activities delivered two times a week for 7 weeks by supportive staff and volunteers trained in CST, on top of their usual care in community centres or residential care homes.
  Interventions: Behavioral: Cognitive Stimulation Therapy
- Usual care group (No Intervention): A total of 64 people with mild-to-moderate cognitive impairment will receive the usual care in community centres or residential care homes.

INTERVENTIONS:
Behavioral: Cognitive Stimulation Therapy — Cognitive stimulation therapy is a non-pharmacological intervention for people with dementia at mild to moderate stages. Group cognitive stimulation therapy is a 14-session intervention delivered twice every week for 7 weeks. In each session, mentally stimulating activities are conducted around a specific themed, such as current affairs, word association, categorising objects, and number game. Each group consists of eight people with similar levels of cognitive impairment, facilitated by two group leaders who lead the activities according to 18 key principles of the therapy, including new associations, opinions rather than facts, implicit learning, and person-centred.
  Arms: CST group

SUMMARY:
This cluster wait-list randomized controlled study investigates the effectiveness of Cognitive Stimulation Therapy (Hong Kong version) delivered by trained supportive staff and volunteers for people in maintaining the quality of life and cognition in people with mild-to-moderate cognitive impairment in community and residential care settings.

DETAILED DESCRIPTION:
Non-pharmacological interventions such as cognitive training, cognitive rehabilitation, and cognitive stimulation aim at slowing down the cognitive decline experienced by a person with dementia. Cognitive stimulation involves a range of group activities and discussions to enhance general cognitive and social functioning. A meta-analysis of 15 studies with a total of 718 persons with dementia showed evidence of benefits of cognitive stimulation on cognitive function, quality of life, and self-reported well-being of the people with dementia . The benefits appeared to add on to medication effects. The clinical improvements in verbal and visual memory, orientation, and auditory comprehension after cognitive stimulation appeared to be able to translate into improvements in real world activity, as seen in enhancement of the communication and social interaction of persons with dementia.

In view of the current evidence, cognitive stimulation is recommended by the National Institute for Health and Clinical Excellence and the Alzheimer's Disease International as an evidence-based, non-pharmacological intervention to be offered to all people with mild-to-moderate dementia. A standard protocol of cognitive stimulation therapy with evidence is a 7-week intervention developed by Spector and her colleagues. It is a series of standardized, well-structured stimulating activities, implemented in a sensitive, respectful and person-centered manner. Group CST typically involves 14 sessions of 45-minute group activities that required cognitive processing delivered over a 7-week period (2 sessions per week, with approximately 45 mins per session). The group size was standardized to be 6 to 8 persons. People with dementia would participate in each of the 14 designated theme activities during each session. The activities aimed at stimulating and engaging persons with dementia in an active way, and providing an optimal learning environment and the positive social benefits of group therapy. Cognitive stimulation therapy can be delivered by non-specialist healthcare workers with minimum training . This allows CST to be used in low-resource environment. Manuals in different languages had been published for the group leaders to follow. Due to this advantage of high reproducibility with high quality evidence support, CST was widely adopted in over 20 countries.

In Hong Kong, there is currently no recommendations or routine provision of cognitive stimulation. In 2015, the standard group CST protocol was culturally adapted for and tested in Chinese people with dementia in Hong Kong (CST-HK). The observed improvements in cognitive outcome was in line with that of overseas studies. The protocol appeared to be feasible and acceptable to Hong Kong Chinese, with high attendance rate (92%) and low attrition rate (13%). Cultural issues identified in the pilot have been published and recommendations were made in adapting the protocol to the Hong Kong cultural settings. A Hong Kong Chinese version of the manual for CST group leaders has been published in 2017.

This study aims to investigate the effectiveness of CST-HK delivered by trained non-professional group leaders in maintaining the quality of life and cognition of people with mild-to-moderate cognitive impairment . As part of project evaluation, it aims to test the effectiveness of CST-HK compared with a wait-list control group who will receive care as usual during the waiting period.

Research Objectives The research aims to investigate the effectiveness of CST-HK among people with mild-to-moderate cognitive impairment in Hong Kong in a larger scale across service settings. It also aims to explore the effectiveness of CST-HK delivered by non-professional staff, as a possible solution to address the shortage of specialized healthcare manpower and increasing demands of non-pharmacological interventions for people with dementia.

Hypotheses The research hypothesized that, compared with the wait-list control group, the group who have received a 7-week (14-session) CST-HK intervention delivered by trained non-professional staff will show greater improvement or maintenance of (1) quality of life; and (2) cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Having a clinical diagnosis of mild-to-moderate dementia, or a cognitive assessment result suggestive of mild-to-moderate cognitive impairment;
* Being able to communicate and understand Cantonese;
* Being able to hear and see well enough to participate in cognitive stimulation activities;
* Having a caregiver who is able to give joint informed consent.

Exclusion Criteria:

* Having major illness(es) that would affect participation (e.g., clinically significant depressive symptoms or psychotic disorders);
* Having behavioural and psychological symptoms (e.g., aggression, inappropriate sexual behaviours, hallucination, delusion) that would interfere with participation in the intervention.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Quality of Life in Alzheimer's Disease | Change from Baseline Quality of Life in Alzheimer's Disease at 8 weeks
  A 13-item scale for self-rating and proxy rating on the quality of life of persons with dementia. The total score ranges from 3 to 52, higher scores means a better outcome.
Alzheimer's Disease Assessment Scale- Cognitive Subscale | Change from Baseline Alzheimer's Disease Assessment Scale- Cognitive Subscale at 8 weeks
  A cognitive function assessment scale for people with dementia covering 11 cognitive domains. The total score ranges from 0 to 70, higher score represents worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hoi Yan Gloria Wong, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Hong Kong Young Women's Christian Association, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguirre E, Woods RT, Spector A, Orrell M. Cognitive stimulation for dementia: a systematic review of the evidence of effectiveness from randomised controlled trials. Ageing Res Rev. 2013 Jan;12(1):253-62. doi: 10.1016/j.arr.2012.07.001. Epub 2012 Aug 7. PMID 22889599
- [Background] Bahar-Fuchs A, Clare L, Woods B. Cognitive training and cognitive rehabilitation for mild to moderate Alzheimer's disease and vascular dementia. Cochrane Database Syst Rev. 2013 Jun 5;2013(6):CD003260. doi: 10.1002/14651858.CD003260.pub2. PMID 23740535
- [Background] Chan IW, Chu LW, Lee PW, Li SW, Yu KK. Effects of cognitive function and depressive mood on the quality of life in Chinese Alzheimer's disease patients in Hong Kong. Geriatr Gerontol Int. 2011 Jan;11(1):69-76. doi: 10.1111/j.1447-0594.2010.00643.x. Epub 2010 Aug 25. PMID 20738410
- [Background] Chu LW, Chiu KC, Hui SL, Yu GK, Tsui WJ, Lee PW. The reliability and validity of the Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog) among the elderly Chinese in Hong Kong. Ann Acad Med Singap. 2000 Jul;29(4):474-85. PMID 11056778
- [Background] Hall L, Orrell M, Stott J, Spector A. Cognitive stimulation therapy (CST): neuropsychological mechanisms of change. Int Psychogeriatr. 2013 Mar;25(3):479-89. doi: 10.1017/S1041610212001822. Epub 2012 Nov 12. PMID 23146408
- [Background] Khan Z, Corbett A, Ballard C. Cognitive stimulation therapy: training, maintenance and implementation in clinical trials. Pragmat Obs Res. 2014 Apr 5;5:15-19. doi: 10.2147/POR.S56000. eCollection 2014. PMID 27774025
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] National Collaborating Centre for Mental Health (UK). Dementia: A NICE-SCIE Guideline on Supporting People With Dementia and Their Carers in Health and Social Care. Leicester (UK): British Psychological Society (UK); 2007. Available from http://www.ncbi.nlm.nih.gov/books/NBK55459/ PMID 21834193
- [Background] Orrell M, Hoe J, Charlesworth G, Russell I, Challis D, Moniz-Cook E, Knapp M, Woods B, Hoare Z, Aguirre E, Toot S, Streater A, Crellin N, Whitaker C, d'Amico F, Rehill A. Support at Home: Interventions to Enhance Life in Dementia (SHIELD) - evidence, development and evaluation of complex interventions. Southampton (UK): NIHR Journals Library; 2017 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK424174/ PMID 28211659
- [Background] Paddick SM. Cognitive stimulation therapy as a low-resource intervention for dementia in sub-saharan africa: Initial results of a controlled trial. Alzheimer's & Dementia: The Journal of the Alzheimer's Association 11(7):607, 2015.
- [Background] Prince M, Bryce R, Ferri C. World Alzheimer Report 2011: The benefits of early diagnosis and intervention. Alzheimer's Disease International (ADI) 2011.
- [Background] Prince M, Wimo A, Guerchet M, Ali G, Wu Y, Prina M. World Alzheimer Report 2015-The Global Impact of Dementia: An analysis of prevalence, incidence, cost and trends. Alzheimer's Disease International (ADI) 2015.
- [Background] Spector A, Orrell M, Woods B. Cognitive Stimulation Therapy (CST): effects on different areas of cognitive function for people with dementia. Int J Geriatr Psychiatry. 2010 Dec;25(12):1253-8. doi: 10.1002/gps.2464. PMID 20069533
- [Background] Spector A, Thorgrimsen L, Woods B, Orrell M. Making a difference: An evidence-based group program to offer cognitive stimulation therapy (CST) to people with dementia; the manual for group leaders (text in chinese). Hong Kong: Hong Kong University Press 2017.
- [Background] Spector A, Thorgrimsen L, Woods B, Royan L, Davies S, Butterworth M, Orrell M. Efficacy of an evidence-based cognitive stimulation therapy programme for people with dementia: randomised controlled trial. Br J Psychiatry. 2003 Sep;183:248-54. doi: 10.1192/bjp.183.3.248. PMID 12948999
- [Background] World Health Organization. Dementia: a public health priority. World Health Organization 2012.
- [Background] Wong GHY, Yek OPL, Zhang AY, Lum TYS, Spector A. Cultural adaptation of cognitive stimulation therapy (CST) for Chinese people with dementia: multicentre pilot study. Int J Geriatr Psychiatry. 2018 Jun;33(6):841-848. doi: 10.1002/gps.4663. Epub 2017 Jan 11. PMID 29717527
- [Background] Woods B, Aguirre E, Spector AE, Orrell M. Cognitive stimulation to improve cognitive functioning in people with dementia. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD005562. doi: 10.1002/14651858.CD005562.pub2. PMID 22336813
- [Background] Yu R, Chau PH, McGhee SM, Cheung WL, Chan KC, Cheung SH, Woo J. Trends in prevalence and mortality of dementia in elderly Hong Kong population: projections, disease burden, and implications for long-term care. Int J Alzheimers Dis. 2012;2012:406852. doi: 10.1155/2012/406852. Epub 2012 Oct 14. PMID 23097740

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT05394584/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT05394584/ICF_001.pdf